CLINICAL TRIAL: NCT01199081
Title: A Randomized, International, Multi-center, Open-label Study to Document Pharmacokinetics and Optimal Timing of Initiation of Dronedarone Treatment Following Long-term Amiodarone in Patients With Paroxysmal or Persistent Atrial Fibrillation Whatever the Reason for the Change of Treatment.
Brief Title: Pharmacokinetics and Optimal Timing of Dronedarone Initiation Following Long-term Amiodarone in Patients With Paroxysmal or Persistent Atrial Fibrillation
Acronym: ARTEMIS AF LT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRONE_C_04629; 2010-019247-19 (EudraCT Number)
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Dronedarone 400 mg twice daily for 8 weeks starting from randomization.
  The last 2 months regimen of Amiodarone 200 mg/day is continued until randomization.
  Interventions: Drug: Dronedarone
- Group B (Experimental): Dronedarone 400 mg twice daily for 6 weeks starting 2 weeks after randomization.
  The last 2 months regimen of Amiodarone 200 mg/day is continued until randomization.
  Interventions: Drug: Dronedarone
- Group C (Experimental): Dronedarone 400 mg twice daily for 4 weeks starting 4 weeks after randomization.
  The last 2 months regimen of Amiodarone 200 mg/day is continued until randomization.
  Interventions: Drug: Dronedarone

INTERVENTIONS:
Drug: Dronedarone — Pharmaceutical form: tablet
  Route of administration: oral (together with meal)
  Dose regimen: 400 mg twice daily
  Other Names: Multaq®; SR33589

SUMMARY:
Primary Objective:

- Explore Dronedarone and active metabolite pharmacokinetic (PK) profiles according to different timings of Dronedarone initiation.

Secondary Objective:

* Explore potential PK interaction between Dronedarone and Amiodarone
* Evaluate the rate of Atrial Fibrillation (AF) recurrence during the study period (from randomization up to 60 days after)
* To assess the safety of the change from Amiodarone to Dronedarone and Dronedarone safety

DETAILED DESCRIPTION:
The maximum study duration per patient is 10 weeks

ELIGIBILITY:
Inclusion criteria:

Screening:

* Paroxysmal or persistent AF having received at least 6 months of amiodarone before screening with at least the last 2 months at a regimen of 200 mg/day (during at least 5 days per week) prior to screening
* Requiring a change from amiodarone treatment whatever the reason, but without liver, lung or thyroid toxicity related to previous use of amiodarone
* At least one cardiovascular risk factor (i.e. age > 70, hypertension, diabetes, prior cerebrovascular disease or left atrial diameter >= 50 mm
* Effective anticoagulation treatments verified by International Normalized Ratio (INR) (target INR > 2)
* QTc Bazett < 500 ms on 12-lead ECG

Randomization:

* Outpatients and Inpatients (except patients hospitalized during screening period for SAE)
* Sinus rhythm
* Effective oral anticoagulation treatment verified by INR (target INR > 2). INR should be closely monitored after initiating dronedarone in patients taking vitamin K antagonist as per their label
* QTc Bazett < 500 ms and PR < 280 ms on 12-lead ECG

Exclusion criteria:

Screening:

* Contraindication to oral anticoagulation
* Acute condition known to cause AF
* Permanent AF
* Bradycardia < 50 bpm at rest on the 12-lead ECG
* History of, or current heart failure or left ventricular systolic dysfunction
* Unstable hemodynamic conditions
* Severe hepatic impairment
* Wolff-Parkinson-White Syndrome
* Previous catheter ablation for atrial fibrillation or catheter ablation scheduled in the next 10 weeks
* Previous history of Amiodarone intolerance or toxicity
* History of thyroid dysfunction
* Mandatory contraindicated concomitant treatment:

  * potent cytochrome P450 (CYP3A4) inhibitors
  * drugs or herbal products that prolong the QT interval and known to increase the risk of Torsade de Pointes
* Previous treatment with class I or class III anti-arrhythmic drugs (including sotalol) other than amiodarone if the anti-arrhythmic drug was taken less than one week before the day of screening (if taken more than one week before screening, the patient can be included)

Randomization

* Bradycardia < 50 bpm on the 12-lead ECG
* History of, or current heart failure or left ventricular systolic dysfunction
* Unstable hemodynamic conditions
* Severe hepatic impairment
* Mandatory contraindicated concomitant treatment:

  * potent cytochrome P450 (CYP3A4) inhibitors
  * drugs or herbal products that prolong the QT interval and known to increase the risk of Torsade de Pointes

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Plasma levels of dronedarone and its metabolite | At randomization (baseline), 3 hours after the first dose of dronedarone, after 1, 2 and 4 weeks of treatment with dronedarone (before dronedarone dose)

SECONDARY OUTCOMES:
Plasma levels of amiodarone and its metabolite | At randomization (baseline), 3 hours after the first dose of dronedarone, after 1, 2 and 4 weeks of treatment with dronedarone (before dronedarone dose)
Number of patients with AF recurrence | From randomization up to 60 days after
Number of patients with Adverse Events of Special Interest (AESIs) | Up to 8 weeks after randomization
  Specific AESIs are: congestive Heart Failure (CHF), Interstitial lung disease , severe skin disorders, peripheral neuropathy including optic neuropathy and increase in alanine aminotransferase (ALT)
Number of patients with symptomatic bradycardia (Heart Rate (HR) < 50 beats per minute at rest) | Up to 8 weeks after randomization
Number of patients with symptomatic tachycardia (HR > 120 beats per minute at rest) | Up to 8 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (40):
- Colombia (6):
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170002, Bucaramanga
  - Investigational Site Number 170003, Cartagena
  - Investigational Site Number 170006, Cartagena
  - Investigational Site Number 170007, Floridablanca
  - Investigational Site Number 170005, Medellín
- Czechia (8):
  - Investigational Site Number 203005, Brno
  - Investigational Site Number 203003, Kladno
  - Investigational Site Number 203002, Olomouc
  - Investigational Site Number 203007, Prachatice
  - Investigational Site Number 203001, Prague
  - Investigational Site Number 203004, Prague
  - Investigational Site Number 203008, Příbram
  - Investigational Site Number 203006, Sternberk
- Denmark (3):
  - Investigational Site Number 208-001, Aarhus
  - Investigational Site Number 208-002, Copenhagen
  - Investigational Site Number 208-003, København S
- France (6):
  - Investigational Site Number 250-004, Amiens
  - Investigational Site Number 250-005, Boulogne-Billancourt
  - Investigational Site Number 250-003, Chambray-lès-Tours
  - Investigational Site Number 250-002, Grenoble
  - Investigational Site Number 250-001, Montpellier
  - Investigational Site Number 250-006, Toulouse
- Germany (5):
  - Investigational Site Number 276-001, Bonn
  - Investigational Site Number 276-002, Chemnitz
  - Investigational Site Number 276-005, Hagen
  - Investigational Site Number 276-003, Nuremberg
  - Investigational Site Number 276-004, Wermsdorf
- Mexico (6):
  - Investigational Site Number 484003, Aguascalientes
  - Investigational Site Number 484002, México
  - Investigational Site Number 484001, San Luis Potosí City
  - Investigational Site Number 484005, San Luis Potosí City
  - Investigational Site Number 484004, Torreón
  - Investigational Site Number 484006, Zapopan
- Spain (6):
  - Investigational Site Number 724004, Barakaldo
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724005, L'Hospitalet de Llobregat
  - Investigational Site Number 724002, Madrid
  - Investigational Site Number 724003, Málaga
  - Investigational Site Number 724006, Valdemoro

REFERENCES:
- [Derived] Naccarelli GV, Bhatt DL, Camm AJ, Le Heuzey JY, Lombardi F, Tamargo J, Martinez JM, Naditch-Brule L; ARTEMIS AF Investigators. Evaluation of the Switch From Amiodarone to Dronedarone in Patients With Atrial Fibrillation: Results of the ARTEMIS AF Studies. J Cardiovasc Pharmacol Ther. 2020 Sep;25(5):425-437. doi: 10.1177/1074248420926874. Epub 2020 Jun 5. PMID 32500725